CLINICAL TRIAL: NCT04998305
Title: A Phase 1/2 Two-center, Double-blind, Randomized, Placebo-controlled Multi-period Crossover (N-of-1) Study to Evaluable the Feasibility, Safety, and Efficacy of TJ-68 in Patients With Amyotrophic Lateral Sclerosis (ALS) and Muscle Cramps
Brief Title: TJ-68 Clinical Trial in Patients With Amyotrophic Lateral Sclerosis (ALS) and Muscle Cramps
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hiroshi Mitsumoto (Other)
Collaborators: Tsumura & Co., Tokyo, Japan (Unknown)
Responsible Party: Sponsor-Investigator, Hiroshi Mitsumoto, Wesley J. Howe Professor of Neurology, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAT0610
Record Dates: First submitted 2021-07-21; First posted 2021-08-10 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Amyotrophic Lateral Sclerosis; Muscle Cramp
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Muscle Cramp | interventions — shakuyaku-kanzoh-toh

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment sequence TJ-68-Placebo-Placebo-TJ-68 (Experimental): Employing an N-of-1, crossover design, each participant in the TJ-68 clinical trial will serve as his/her control. The participation will last for 11 weeks - four, 2-week treatment periods with 1-week washout (WO) period between each treatment period. Participants (n=13) will be randomized to the following treatment sequences:
  TJ-68, placebo, placebo, TJ-68 (1 week WO between each treatment period)
  Interventions: Drug: TJ-68; Drug: Placebo
- Treatment sequence Placebo-TJ-68-TJ-68-Placebo (Experimental): Employing an N-of-1, crossover design, each participant in the TJ-68 clinical trial will serve as his/her control. The participation will last for 11 weeks - four, 2-week treatment periods with 1-week washout (WO) period between each treatment period. Participants (n=13) will be randomized to the following treatment sequences:
  placebo, TJ-68, TJ-68, placebo (1 week WO between each treatment period)
  Interventions: Drug: TJ-68; Drug: Placebo

INTERVENTIONS:
Drug: TJ-68 — For two periods (one period = 2 weeks) during the 11-week participation, participants will take 2.5 g of TJ-68 for three times per day before meals. It will be administered by dissolving 2.5 g of TJ-68 powder in 1 oz. of lukewarm water.
  Other Names: Shakuyakukanzoto
Drug: Placebo — For two periods (one period = 2 weeks) during the 11-week participation, participants will take 2.5 g of placebo for three times per day before meals. It will be administered by dissolving 2.5 g of the placebo powder in 1 oz. of lukewarm water.
  Other Names: Placebo Tablet

SUMMARY:
The primary objective of the study is to demonstrate the safety and potential efficacy of TJ-68 for improving muscle cramps in participants with ALS based on a two-site, randomized, placebo-controlled double-blind multi-period crossover (N-of-1) study design.

DETAILED DESCRIPTION:
In Japan, TJ-68 is a common Kampo medicine prescribed by Japanese physicians to manage muscle cramps or pain of diverse origins. In the USA, there are no effective medications to control muscle cramps and no approved medications to specifically treat muscle cramps. Quinine sulfate and Mexiletine have shown some effect with additional safety considerations. The fact that TJ-68 has been commonly used for the treatment of muscle cramps in Japan and the lack of available medications for cramps in ALS represent the fundamental rationale for this proposal.

This is a phase 1/2, two-site, double-blinded, randomized, placebo-controlled, multi-period crossover clinical trial for individuals with ALS and muscle cramps. Participants will be enrolled in the study for 11 weeks and receive TJ-68, also known as Shakuyakukanzoto - a kampo, herbal medicine - to assess its effect in relieving muscle cramps. This clinical trial employs N-of-1 study design in which all participants will receive TJ-68 and placebo at certain points, serving as their own controls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ALS, PMA or PLS based on the El Escorial ALS Diagnostic Criteria or based on more recently revised Gold Coast ALS diagnostic criteria
* Experiences at least one muscle cramp in any muscle per day
* Age 20 to 84 years old
* Forced vital capacity is 45% of normal or greater in a seated position
* Able to swallow liquid via the mouth or be given via a feeding tube
* Caregiver available to assist with speaking or writing on behalf of the participant if they are not able to speak or write due to the disease
* Able to comprehend and willing to give (sign) the informed consent
* Willing to commute to the study site for the frequent visits, including a screening visit (study visits at the end of week 2, 5, 8 and 11)
* Taking a stable dose of Riluzole (Rilutek), Edaravone (Radicava), and/or sodium phenylbutyrate/taurursodiol (Relyvrio) for at least a month before randomization and not expected to require dose titration or initiation of these medications during the study period
* Willing to discontinue over-the-counter (OTC) products containing any peony root, Glycyrrhiza, or both
* Willing to discontinue Mexiletine, Quinine sulfate, or Ranolazine during the study period
* Willing to avoid food, beverages, and medications that may induce or inhibit metabolism of enzyme of transporters.
* Willing to refrain from initiation or dose adjustment of baclofen, gabapentin, pregabalin, and/or memantine during the study period (stable dosing of these medications is allowed).
* Willing to practice contraceptive measures for male and female patients.

Exclusion Criteria:

* History of allergic reactions to peony root, Glycyrrhiza, or FD&C Yellow No. 5 (tartrazine)
* Takes any medication known to increase the risk of pseudoaldosteronism or hypokalemia, including corticosteroids and diuretics (except potassium sparing diuretics, such as spironolactone or amiloride)
* History of pseudoaldosteronism or hypokalemia or current use of potassium supplementation
* Screening potassium level 3.4 mEq/L or less
* Screening diastolic blood pressure (DBP) more than 90 mmHg or systolic blood pressure (SBP) more than 150 mmHg after sufficient rest
* Screening albumin below normal laboratory level either at the Columbia or Mayo Clinic laboratory
* Screening bicarbonate or carbon dioxide level less than 29 mmol/L, suggesting metabolic alkalosis
* Screening sodium level greater than 145 mmol/L, suggesting hypernatremia
* Unstable or active medical or neurological (other than ALS) diseases which require treatment
* Failure of Capacity Assessment
* Not able and/or willing to comprehend and sign the informed consent
* Not able to speak or write English to complete the primary outcome measure, MCS
* Taking any experimental medication or unapproved medications directed at treating muscle cramps
* Those who are pregnant or breast feeding
* Those who have renal or hepatic impairment

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Mistumoto, MD, Dsc., Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitsumoto H, Cheung K, Oskarsson B, Andrews HF, Jang GE, Andrews JA, Shah JS, Fernandes JA, McElhiney M, Santella RM. Randomized double-blind personalized N-of-1 clinical trial to test the safety and potential efficacy of TJ-68 for treating muscle cramps in amyotrophic lateral sclerosis (ALS): study protocol for a TJ-68 trial. Trials. 2023 Jul 10;24(1):449. doi: 10.1186/s13063-023-07424-8. PMID 37430314

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence TJ-68-Placebo-Placebo-TJ-68: Employing an N-of-1, crossover design, each participant in the TJ-68 clinical trial will serve as his/her control. The participation will last for 11 weeks: four 2-week treatment periods with 1-week washout (WO) period between each treatment period. Participants will be randomized to the following treatment sequences:
  TJ-68, placebo, placebo, TJ-68 (1 week WO between each treatment period)
- Treatment Sequence Placebo-TJ-68-TJ-68-Placebo: Employing an N-of-1, crossover design, each participant in the TJ-68 clinical trial will serve as his/her control. The participation will last for 11 weeks: four 2-week treatment periods with 1-week washout (WO) period between each treatment period. Participants will be randomized to the following treatment sequences:
  placebo, TJ-68, TJ-68, placebo (1 week WO between each treatment period)
Period: Treatment (2 Weeks)
Arm/Group | Treatment Sequence TJ-68-Placebo-Placebo-TJ-68 | Treatment Sequence Placebo-TJ-68-TJ-68-Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Treatment Sequence TJ-68-Placebo-Placebo-TJ-68 | Treatment Sequence Placebo-TJ-68-TJ-68-Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Treatment (2 Weeks)
Arm/Group | Treatment Sequence TJ-68-Placebo-Placebo-TJ-68 | Treatment Sequence Placebo-TJ-68-TJ-68-Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Treatment Sequence TJ-68-Placebo-Placebo-TJ-68 | Treatment Sequence Placebo-TJ-68-TJ-68-Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Treatment (2 Weeks)
Arm/Group | Treatment Sequence TJ-68-Placebo-Placebo-TJ-68 | Treatment Sequence Placebo-TJ-68-TJ-68-Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Treatment Sequence TJ-68-Placebo-Placebo-TJ-68 | Treatment Sequence Placebo-TJ-68-TJ-68-Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Treatment (2 Weeks)
Arm/Group | Treatment Sequence TJ-68-Placebo-Placebo-TJ-68 | Treatment Sequence Placebo-TJ-68-TJ-68-Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence TJ-68-Placebo-Placebo-TJ-68 | Treatment Sequence Placebo-TJ-68-TJ-68-Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8.15) | 62.8 (7.29) | 62.9 (7.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (MCS-VAS) Score
Description: This is designed to measure improvements in muscle cramps. MCS-VAS indicates the level to which muscle cramps affect overall daily activity. The score ranges from 0 to 10; 0 indicates no interference and 10 indicates severe interference with overall daily activity. MCS-VAS will be administered by a trained evaluator to reduce recall bias and lack of insight, which can limit subjective assessments. To minimize carryover effects, results reflect the average of the scores taken at the second week of each treatment period.
Time Frame: Assessed at Baseline, Week 2, Week 5, Week 8 and Week 11; Week 2 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Participants who were administered the placebo during the first 2-week treatment period.
- TJ-68: Participants who were administered TJ-68 during the first 2-week treatment period.
Arm/Group | Placebo | TJ-68
Number analyzed (Participants) | 11 | 11
score on a scale | 2.07 (2.03) | 1.7 (1.91)

2. Secondary Outcome: Overall Muscle Cramp Scale (MCS) Score
Description: Changes in trigger, frequency, severity, and location of muscle cramps will be measured by administering all of MCS questions. Motor behaviors which trigger muscle cramps and muscle cramps' effects on sleep quality will also be measured. The score for each component of MCS -- trigger, frequency, severity, location, behavior, and effect on sleep quality -- will range from 1 to 5, with the severity increasing from 1 to 5. The total score range is 6 to 30. All of the MCS components will be administered by a trained evaluator and evaluated by the investigator. To minimize carryover effects, results reflect the average of the scores taken at the second week of each treatment period.
Time Frame: Assessed at Baseline, Week 2, Week 5, Week 8 and Week 11; Week 2 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TJ-68
Number analyzed (Participants) | 11 | 11
score on a scale | 14.7 (5.07) | 13.1 (5.81)

3. Secondary Outcome: Self-reported Cramp Pain Score
Description: Cramp pain will be measured on a scale of 0 to 10 with 0 indicating no pain and 10 indicating severe pain. To minimize carryover effects, results reflect the average of the scores taken at the second week of each treatment period.
Time Frame: Assessed at Baseline, Week 2, Week 5, Week 8 and Week 11; Week 2 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TJ-68
Number analyzed (Participants) | 11 | 11
score on a scale | 0.59 (0.41) | 0.49 (0.46)

4. Secondary Outcome: ALSFRS-R Score
Description: Changes in functionality due to disease progression will be measured by administering ALSFRS-R to participants. ALSFRS-R includes 12 questions that can have a score of 0 to 4. A score of 0 on a question would indicate no function while a score of 4 would indicate full function. Total score range is 0 to 48. To minimize carryover effects, results reflect the average of the scores taken at the second week of each treatment period.
Time Frame: Assessed at Baseline, Week 2, Week 5, Week 8 and Week 11; Week 2 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TJ-68
Number analyzed (Participants) | 11 | 11
score on a scale | 34.1 (5.37) | 34.5 (5.39)

5. Secondary Outcome: Clinical Global Impression of Changes (CGIC) Score
Description: Changes in participant's feelings since the start of dosing will be measured by using a score of 1 to 7 with 1 indicating "very much improved" and 7 indicating "very much worse." To minimize carryover effects, results reflect the average of the scores taken at the second week of each treatment period.
Time Frame: Assessed at Baseline, Week 2, Week 5, Week 8 and Week 11; Week 2 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TJ-68
Number analyzed (Participants) | 11 | 11
score on a scale | 3.48 (1.24) | 2.95 (1.28)

6. Secondary Outcome: ALSAQ-5 (Quality of Life Questionnaire) Score
Description: Participants' motor functions and resulting quality of life will be measured by asking questions about their ability to perform certain tasks or feelings of hopelessness within the last two weeks. Participants can answer by saying never, rarely, sometimes, often, or always/cannot do at all. The ALSAQ-5 full score range is from 0 to 100, with 0 reflecting the best health state. To minimize carryover effects, results reflect the average of the scores taken at the second week of each treatment period.
Time Frame: Assessed at Baseline, Week 2, Week 5, Week 8 and Week 11; Week 2 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TJ-68
Number analyzed (Participants) | 11 | 11
score on a scale | 4.83 (2.39) | 5 (3.05)

7. Secondary Outcome: Goal Attainment Scale (GAS) Score
Description: Participant and the evaluator will collaborate and establish a goal. Progression of goal achievement will be measured over the course of participation and scored from -2 to +2 with -2 indicating "(achievement) much worse than expected" and +2 indicating "(achievement) much better than expected." To minimize carryover effects, results reflect the average of the scores taken at the second week of each treatment period.
Time Frame: Assessed at Baseline, Week 2, Week 5, Week 8 and Week 11; Week 2 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TJ-68
Number analyzed (Participants) | 11 | 11
score on a scale | 0.50 (1.14) | 0.67 (1.11)

ADVERSE EVENTS:
Time Frame: 11 weeks
Arm/Group | Placebo | TJ-68
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 2/11
Other Adverse Events (participants affected / at risk) | 3/11 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | TJ-68 (N=11)
Respiratory distress due to RSV (Infections and infestations) | 0 | 1
Diverticulitis with pericecal abscess (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | TJ-68 (N=11)
Facial rash (General disorders) | 0 | 1
Abdominal bloating (Gastrointestinal disorders) | 0 | 1
Stomachache (Gastrointestinal disorders) | 0 | 1
Elevated blood pressure (General disorders) | 0 | 1
Flu-like symptoms (General disorders) | 1 | 1
Joint pain (General disorders) | 0 | 1
Scleral erythema (Eye disorders) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Fatigue (General disorders) | 1 | 0
Sinusitis (General disorders) | 1 | 0
Hypertension (General disorders) | 1 | 0
Fall (General disorders) | 1 | 0
Hypokalemia (Blood and lymphatic system disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT04998305/Prot_SAP_000.pdf